CLINICAL TRIAL: NCT06155812
Title: Simultaneous Administration of Norepinephrine, Angiotensin II, and Vasopressin in Septic Shock Patients
Brief Title: Multimodal Vasopressor Strategy in Septic Shock
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Ziga Kalamar, Principal Investigator, University Medical Centre Maribor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRP-2023/01-03
Record Dates: First submitted 2023-11-09; First posted 2023-12-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Shock, Septic
Keywords: Vasopressor agents; Angiotensin II; Vasopressin; Norepinephrine; Renin; Lactate
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus

STUDY DESIGN:
Intervention Model Description: Vasopressors will be administered successively in the control group. In the experimental group norepinephrine, angiotensin II, and vasopressin will be administered simultaneously.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STEPWISE VASOPRESSOR SEPTIC SHOCK MANAGEMENT (Active Comparator): Regimen: Norepinephrine increases of 0.05-0.1 mcg/kg/min up to 0.5 mcg/kg/min, followed by vasopressin (administered at a fixed dose of 0.03 IE/min). If MAP remains < 65 mmHg, norepinephrine will be titrated above dose of 0.5 mcg/kg/min until MAP ≥ 65 mmHg. Maximum norepinephrine dose as per clinical team decision. Initiation of additional vasoactive drugs (epinephrine, Ang II methylene blue or dopamine) as per clinical team decision. Initiation of inotropes (dobutamin, levosimendan, milrinone) as per clinical team decision.
  Interventions: Other: Successive administration of vasopressors
- BALANCED MULTIMODAL VASOPRESSOR SEPTIC SHOCK MANAGEMENT (Experimental): Regimen: Simultaneous administration of norepinephrine, angiotensin II and vasopressin at equivalent starting doses (equivalent to approximately 0.05 mcg/kg/min of norepinephrine). Increments of 0.05 mcg/kg/min of equivalent doses of all three vasopressors every 3-5 min until MAP ≥ 65 mmHg is reached (vasopressin will be administered at a maximum dose of 0.03 IE/min, AT II will be administered at a maximum dose of 100 ng/kg/min). Initiation of additional vasoactive drugs (epinephrine, methylene blue or dopamine) as per clinical team decision. Initiation of inotropes (dobutamin, levosimendan, milrinone) as per clinical team decision.
  Interventions: Other: Simultaneous administration of vasopressors

INTERVENTIONS:
Other: Simultaneous administration of vasopressors — Early, simultaneous administration of norepinephrine, angiotensin II, and vasopressin.
  Arms: BALANCED MULTIMODAL VASOPRESSOR SEPTIC SHOCK MANAGEMENT
Other: Successive administration of vasopressors — Administration and titration of norepinephrine and vasopressin. Administration of additional vasoactive drugs (epinephrine, methylene blue, angiotensin II or dopamine) as per clinical team. Initiation of inotropes (dobutamin, levosimendan, milrinone) as per clinical team decision.
  Arms: STEPWISE VASOPRESSOR SEPTIC SHOCK MANAGEMENT

SUMMARY:
The goal of this prospective randomized controlled trial is to compare the effects of classic stepwise vs. early balanced multimodal vasopressor strategies in septic shock.

DETAILED DESCRIPTION:
CONTROL GROUP(Classic stepwise vasopressor administration):

Patients will be started on norepinephrine with increases of 0.05-0.1 mcg/kg/min up to 0.5 mcg/kg/min, followed by vasopressin (administered at a fixed dose of 0.03 IE/min). If MAP remains < 65 mmHg, norepinephrine will be titrated above dose of 0.5 mcg/kg/min until MAP ≥ 65 mmHg. Initiation of additional vasoactive drugs (epinephrine, Ang II, methylene blue or dopamine) as per clinical team decision. Initiation of inotropes (dobutamine, milrinone, levosimendan) as per clinical team decision.

EXPERIMENTAL GROUP(Balanced multimodal vasopressor administration):

Early, simultaneous start of norepinephrine, angiotensin II and vasopressin at equivalent starting doses (equivalent to approximately 0.05 mcg/kg/min of norepinephrine). Increments of 0.05 mcg/kg/min of equivalent doses of all three vasopressors every 3-5 min until MAP ≥ 65 mmHg is reached (vasopressin will be administered at a maximum dose of 0.03 IE/min, Ang II will be administered at maximum dose of 100ng/kg/min). Initiation of additional vasoactive drugs (epinephrine, methylene blue or dopamine) as per clinical team decision. Initiation of inotropes (dobutamine, milrinone, levosimendan) as per clinical team decision.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years).
* Sepsis (an acute change in total Sequential Organ Failure Assessment (SOFA) score ≥2 points consequent to infection) with persisting hypotension requiring vasopressors to maintain MAP ≥65 mm Hg and having a serum lactate level >2 mmol/L despite adequate volume resuscitation (20-30ml/kg in 3 hours).
* Vasopressor requirement of ≥0,15 μg/kg/min equivalent of norepinephrine base.
* Patients are required to have central venous access and an arterial line present, and these are expected to remain present for at least the initial 72 hours of study.
* Patients are required to have an urinary catheter present, and it is expected to remain present for at least the initial 72 hours of study.
* Patients must have cardiac index (CI) >2.3 L/min/m2 (measured by bedside echocardiography, pulse contour cardiac output (PiCCO) or Swan-Ganz catheter).

Exclusion Criteria:

* Death expected <24 hours.
* Pregnancy (suspected or confirmed).
* Surgery expected for source of infection.
* Inter-hospital transfer expected during first 72 hours of hospitalization.
* Liver failure with a Model for End-Stage Liver Disease (MELD) score of ≥30.
* Patients with acute mesenteric ischemia or a history of mesenteric ischemic.
* Patients with Raynaud's phenomenon, systemic sclerosis or vasospastic disease.
* Patients with active bleeding and an anticipated need (within 48 hours of initiation of the study) for transfusion of >4 units of packed red blood cells.
* Patients with a known allergy to mannitol.
* Patients on veno-arterial (VA) ECMO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Rate of change in renin levels | 72 hours
  There is an increasing amount of data that renin is the best marker of tissue hypoperfusion and predictor of ICU mortality in patients with sepsis and septic shock, even outperforming lactate. Renin increased between the first and third day in non-survivors, but dropped in survivors. The rate of change in renin concentration but not lactate concentration in ICU patients over first 72 hours is associated with in hospital mortality.

SECONDARY OUTCOMES:
Compare lactate levels | 72h
  In critically ill patients, plasma lactate is commonly used to guide hemodynamic resuscitation. Hyperlactatemia has been widely recognized as a marker of tissue hypoxia/hypoperfusion but it can also result from increased or accelerated aerobic glycolysis during the stress response and may represent an important energy source in critically ill patients. Resuscitation to normalize lactate levels could worsen physiological status.
Compare Δ Sequential Organ Failure Assessment (SOFA) score | 72 hours
  The purpose is to monitor the rate of organ dysfunction. Score ranges from 0 (best) to 24 (worst) points.
Compare acute kidney injury rate | 72 hours
  The purpose is to monitor acute kidney injury based on Improving Global Outcomes (KDIGO) definition and staging system.

OTHER OUTCOMES:
Survival to ICU discharge | From date of ICU admission until date of ICU discharge or death during ICU stay whichever came first, assessed up to 8 weeks
28-day mortality | 28 days after first admission to the ICU
Renal replacement therapy requirement during ICU stay. | From date of ICU admission until date of ICU discharge or death during ICU stay whichever came first, assessed up to 8 weeks
Vasopressor cumulative dose requirement. | 72 hours
Quality of life assessment 90 days after ICU admission (using EQ-5D standardized questionnaire). | 90 days after ICU admission if alive

CONTACTS AND LOCATIONS:
Overall Officials: Žiga Kalamar, MD, Principal Investigator — University Medical Centre Maribor
Locations (2):
- University Hospital Centre Zagreb, Zagreb, Croatia
- Medical intensive care unit UMC Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: After November 2026

REFERENCES:
- [Derived] Kalamar Z, Gorenjak M, Landoni G, Markota A. Early multimodal vasopressor strategy in septic shock (TRICYCLE)-Study protocol for a randomized controlled clinical trial. PLoS One. 2025 Aug 29;20(8):e0331304. doi: 10.1371/journal.pone.0331304. eCollection 2025. PMID 40880376